CLINICAL TRIAL: NCT03988283
Title: A Pilot Study to Assess the Safety, Feasibility, and Preliminary Efficacy of a Neoepitope-based Personalized DNA Vaccine Approach in Pediatric Patients With Recurrent Central Nervous System Tumors
Brief Title: Neoepitope-based Personalized DNA Vaccine Approach in Pediatric Patients With Recurrent Central Nervous System Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Children's Discovery Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202211187
Record Dates: First submitted 2019-06-12; First posted 2019-06-17 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Pediatric Recurrent Central Nervous System Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Personalized neoantigen DNA vaccine (Experimental): Patients will receive the vaccine monthly (+/- 3 days) for 6 doses as a priming phase followed by booster injections quarterly Q3mo thereafter. If sufficient quantities of vaccine are available, vaccination may continue until development of intolerance or disease progression in the case of fatal high grade neoplasms or for up to one year. Additionally, patients with non-fatal tumors who complete one year of vaccinations and have stable disease at the completion of treatment will be given the option of resuming vaccinations if they develop subsequent progression.
  Interventions: Biological: Personalized neoantigen DNA vaccine; Device: Papivax Biotech TDS-IM v2.0; Procedure: Peripheral blood draw

INTERVENTIONS:
Biological: Personalized neoantigen DNA vaccine — At each vaccination time point, patients will receive one injection of the neoantigen DNA vaccine, one injection into the vastus lateralis.
Device: Papivax Biotech TDS-IM v2.0 — All study injections will be given intramuscularly using an integrated electroporation device (TDS-IM v2.0 device - Papivax Biotech).
Procedure: Peripheral blood draw — -After trial enrollment and up to 7 days after the first vaccine dose (baseline); no more than 2 weeks after the 3rd vaccine dose; no more than 2 weeks after the 6th vaccine dose; two weeks after the last dose; time of progression or discontinuation (optional)

SUMMARY:
The purpose of this research study is to learn about the safety and feasibility of giving a personalized DNA vaccine to people with central nervous system tumors that have returned or have been resistant to treatment.

ELIGIBILITY:
Step 1 Eligibility Criteria for Tissue Sequencing

Inclusion Criteria:

* Any patient between the ages of 12 and 25 years of age (inclusive) who was diagnosed with a pediatric CNS (brain or spine) of any histologic subtype, who has now developed recurrent or refractory disease.
* All patients enrolled in this trial will receive treatment for recurrent and/or refractory pediatric CNS tumors, including systemic agents, investigational agents, or radiation therapy, prior to receiving the neoantigen DNA vaccine. Co-enrollment to another interventional clinical trial is permitted during the vaccine manufacture period.
* Availability of tissue collected after progression for sequencing to determine presence of targetable neoantigen. This may be fresh tissue collected as part of routine care, another research project or banked fresh frozen samples from tissue obtained at the time of progression from a biopsy, subtotal resection, total gross resection, or re-resection.
* Life expectancy > 24 weeks.
* Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable) or patient has a guardian who has the ability to understand and willingness to sign an IRB approved written informed consent document.
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, or should a man suspect he has fathered a child, s/he must inform her treating physician immediately.

Step 1 Exclusion Criteria:

* A history of other malignancy ≤ 3 years previous with the exception of non-melanoma skin cancer, any in situ cancer that has been successfully resected and cured, treated superficial bladder cancer, or any early-stage solid tumor that was successfully resected without need for adjuvant radiation or chemotherapy.
* Known allergy, or history of serious adverse reaction to, vaccines such as anaphylaxis, hives, or respiratory difficulty.
* Uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* History of immunodeficiency disorder or autoimmune condition requiring active immunosuppressive therapy. This includes inflammatory bowel disease, ulcerative colitis, Crohn's disease, systemic vasculitis, scleroderma, psoriasis, multiple sclerosis, hemolytic anemia, immune-mediated thrombocytopenia, rheumatoid arthritis, systemic lupus erythematosus, Sjögren's syndrome, sarcoidosis, or other rheumatologic disease or any other medical condition or use of medication which might make it difficult for the patient to complete the full course of treatments or to generate an immune response to vaccines.
* Patients with HIV are eligible unless their CD4+ T-cell counts are < 350 cells/mcL or they have a history of AIDS-defining opportunistic infection within the 12 months prior to registration. Concurrent treatment with effective ART according to DHHS treatment guidelines is recommended.
* Presence of clinically significant increased intracranial pressure (e.g. impending herniation) or hemorrhage, uncontrolled seizures, or requirement for immediate palliative treatment.
* Individuals in whom a measurement of the circumference of the thigh at the midpoint between the hip and knee is < 35 cm.
* Individuals in whom a skinfold measurement of the cutaneous and subcutaneous tissue for eligible injection sites (left and right vastus laterals muscles) exceeds 50 mm.
* Individuals in whom the ability to observe possible local reactions at the eligible injection sites is, in the opinion of the investigator, unacceptably obscured due to a physical condition (e.g. hypertrophic skin patches, keloids, or other conditions which could interfere with the administration procedure or subsequent assessment of local reactogenicity) or permanent body art.
* Has a metal implant or implantable device within the area of the electroporation injection or has any non-removable electronic stimulation device, such as cardiac demand pacemaker, automatic implantable cardiac defibrillator, nerve stimulator, or deep brain stimulator.
* Acute or chronic, clinically significant hematologic, pulmonary, cardiovascular, or hepatic or renal functional abnormality as determined by the investigator based on medical history, physical examination, EKG, and/or laboratory screening test.
* Any chronic or active neurologic disorder, including seizures and epilepsy, excluding a single febrile seizure as a child.

Step 2 Eligibility Criteria for Treatment Administration

Inclusion Criteria:

* Personalized neoantigen DNA vaccine manufactured for administration.
* Karnofsky/Lansky performance status ≥ 60%
* Life expectancy > 12 weeks.
* Prior therapy washout requirements (with exception of bevacizumab):

  * Myelosuppressive chemotherapy: Participants must have received their last dose of known myelosuppressive anticancer chemotherapy at least 3 weeks prior to first dose of vaccine or at least 6 weeks prior if nitrosurea.
  * Biologic agent: Participant must have received their last dose of the biologic agent at least 7 days prior to first dose of vaccine.

    * For agents that have known adverse events occurring beyond 7 days after administration, this period must be extended to beyond the time during which adverse events are known to occur. The duration of this interval should be discussed with the study PI.
    * For biologic agents that have a prolonged half-life, the appropriate interval since last treatment should be discussed with the PI prior to first dose of vaccine.
  * Monoclonal antibody treatment: At least three half-lives must have elapsed prior to first dose of vaccine. Such participants should be discussed with the PI prior.
  * Bone Marrow Transplant: Participant must be:

    * ≥ 6 months since allogeneic bone marrow transplant prior to first dose of vaccine.
    * ≥ 3 months since autologous bone marrow/stem cell prior to first dose of vaccine.
  * Radiotherapy (in instances of lesions amenable to radiotherapy, such as bone metastases or metastases causing nerve impingement): The last fraction must have been at least 4 weeks prior to first dose of vaccine.
  * Investigational agents: The last dose must have been at least 4 weeks prior to first dose of vaccine.
* Adequate bone marrow and organ function as defined below:

  * Absolute neutrophil count ≥ 1.5 K/cumm
  * Platelets ≥ 100 K/cumm
  * Hemoglobin level ≥ 8 g/dL
  * Total bilirubin ≤ 1.5 x institutional upper limit of normal (IULN)
  * AST(SGOT)/ALT(SGPT) ≤ 3.0 x IULN
  * Creatinine ≤ IULN OR creatinine clearance ≥ 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Any adverse event patients may have experienced during prior therapy must have resolved to ≤ grade 1 CTCAE v5.
* Systemic corticosteroid therapy is permitted provided dosing is minimal based on age, defined as 0.1mg/kg/day with a max of 4mg daily (dexamethasone or equivalent) on the day of vaccine administration. Participants using topical, ocular, intra-articular, or intranasal/inhaled steroids may participate. Brief courses of corticosteroids for prophylaxis (eg, contrast dye allergy) or study treatment-related standard premedication are permitted.
* Bevacizumab will be allowed if given for symptomatic control of vasogenic edema and to avoid high dose of corticosteroids.

Step 2 Exclusion Criteria:

* No candidate neoantigen identified during the vaccine evaluation process.
* Ongoing or active infection requiring systemic therapy (e.g. active HBV or HCV infection that requires treatment) or causing fever (temperature > 38.1˚C) or subjects with unexplained fever (temperature > 38.1˚C) within 7 days prior to the first vaccine dose.
* Administration of live vaccine within 30 days prior to first dose of vaccine. Participants may receive the COVID-19 vaccine within this time period as it is not a live vaccine.
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative pregnancy test within 7 days of first dose of vaccine.
* Syncopal episode within 12 months of first dose of vaccine.

Max Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 7 (Estimated)
Dates: Start 2024-10-02 (Actual); Primary Completion 2029-03-31 (Estimated); Study Completion 2031-02-28 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of adjuvant personalized neoantigen DNA vaccine as measured by the number of grade 3 and 4 adverse events | Through 30 days after completion of treatment (estimated to be 13 months)
Feasibility of adjuvant personalized neoantigen DNA vaccine as measured the number of participants that had a neoantigen-specific DNA vaccine generated | From time of resection to time of initiation (approximately 12-14 weeks)

SECONDARY OUTCOMES:
Median Progression Free Survival (PFS) | 2 years
  * PFS is defined as the duration of time from date of first dose of vaccine to date of progression or evidence of last progression free time.
  * Progressive Disease (PD): At least a 25% increase in the sum of products of perpendicular diameters of at least 1 target lesion, taking as reference the smallest sum of products of perpendicular diameters on study (this includes the baseline sum if that is the smallest on study). The absolute increase in any dimension must be at least 5mm when calculating the products of perpendicular diameters. Appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions on stable or increasing doses of corticosteroids compared with baseline scan or best response after initiation of therapy* not caused by comorbid events.
Median Overall Survival | 2 years
  -OS is defined as date of first dose of vaccine to date of death or date of last known alive.

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Huang, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu